CLINICAL TRIAL: NCT01945684
Title: A Randomized, Double Blind, Multi-center, Active Drug Controlled, Phase III Clinical Trial to Compare the Safety and Efficacy of DWP450 Versus Botox® in Treatment of Post Stroke Upper Limb Spasticity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DW_DWP450002
Record Dates: First submitted 2013-09-16; First posted 2013-09-18 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-03

CONDITIONS: Spasticity; Stroke
MeSH Terms: conditions — Muscle Spasticity; Stroke | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin type A (DWP450) (Experimental): DWP450: Botulinum toxin type A
  Interventions: Drug: Botulinum toxin type A
- Botulinum toxin type A (Botox®) (Active Comparator): Botox®: Botulinum toxin type A
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Maximum dose 360 U
  Other Names: Assigned Interventions; Experimental: DWP450; Botulinum toxin type A Drug: Botulinum toxin type A; Active Comparator: Botox®; Botulinum Toxin type A Drug: Botulinum Toxin type A (Botox®)

SUMMARY:
Purpose: This study is a Randomized, Double Blind, Multi-center, Active Drug Controlled, Phase III Clinical Trial to Compare the Safety and Efficacy of DWP450 Versus Botox® in Treatment of Post Stroke Upper Limb(wrist, finger, elbow, thumb)Spasticity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult patients
2. ≥ 6 weeks since the last stroke

Exclusion Criteria:

1.Patients with diagnosed neuromuscular disorders such as Lamber-Eaton syndrome, myasthenia gravis, or amyotrophic lateral sclerosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2013-09; Primary Completion 2014-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
The change in MAS(Modified Ashworth Scale)grade for Wrist flexor | at 4 week
  The change in MAS (Modified Ashworth Scale) grade from baseline at week 4 for wrist flexor muscle tone

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, 41, Borame-Gill, Dong Gjak-Gu, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No